CLINICAL TRIAL: NCT06618339
Title: Randomized Controlled Trials to Measure Neurophysiological Effects Using EEG Signals, Artificial Intelligence and Neuropsychological Techniques of a Mindfulness-Based Intervention in Young Adults with Symptoms of Anxiety and Depression
Brief Title: Clinical Trials to Evaluate Neurophysiological and Neuropsychological Effects of a Mindfulness-based Intervention
Acronym: PRESENTE-IA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Gilberto Galindo, Full time Professor, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 215/2/C/63/24
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Anxiety Depression (Mild or Not Persistent)
Keywords: Anxiety; Depression
MeSH Terms: conditions — Lymphoma, Follicular; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychoeducation (Other): 8 session Psychoeducation, for anxiety and depression.
  Interventions: Behavioral: Mindfulness-based intervention
- Cognitive flexibility and resilence (Sham Comparator): 8 Session cognitive flexibility and resilience trainning.
  Interventions: Behavioral: Mindfulness-based intervention

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — 8 Session Mindfulness-based intervention

SUMMARY:
Depression and anxiety are conditions with a high prevalence in the world population and youth are no exception. In developing countries it is reported that given the conditions of social disadvantage, anxiety and depression are higher, resulting in compromised psychological well-being and mental health. Therefore, treatments that help in the care and prevention of these disorders from youth are important. In the case of contemporary psychology, Mindfulness treatments have emerged as an alternative treatment for some of the symptoms of depression, anxiety and emotional discomfort, showing evidence of increased improvement in the overall quality of life. The project responds to global mental health demands and will provide the institution, as well as external collaborating institutions and society in general, with guidelines to carry out brief and effective interventions for these problems and will develop clinical evidence and technological tools for their analysis. Objective: To compare the neurophysiological effects by means of EEG signals and machine learning or deep learning techniques and neuropsychological effects of a brief treatment based on mindfulness-based intervention techniques as an alternative intervention for the reduction of anxiety and depression symptoms against the effects of psychoeducation groups and placebo group in young adults. Methodology: Factorial design of cases and controls according to the guidelines for randomized controlled trials CONSORT. Participants (n=125) will be randomized triple-blinded with neuropsychological and neurophysiological assessments. The results of the project will generate basic evidence on the condition of brain functioning at the neurophysiological level, its performance to perform processes of utmost relevance to solve daily life problems and psychological well-being, as well as support the development of techniques for specialists in behavioral analysis and mental health and engineering sciences for the creation and implementation of programs and strategies for the prevention, identification, care and evaluation of mental health and social well-being, with a scientific and community health approach.

DETAILED DESCRIPTION:
Protocol

Study type. Factorial case-control design according to the guidelines for CONSORT randomized controlled trials (Cuschieri, 2019). Participants will be randomized triple-blinded.

Stage 1. Clinical Trials Registration. Involvement Participant eligibility assessments (n = 125). Participant permanence analysis, inclusion and exclusion criteria. Randomized groups (n = 125) Blinded 1 Group assignment A = placebo treatment control group, B = mindfulness-based intervention group, C = PE-based intervention group.

Randomization of participants to the intervention Blind 2 Group 1: A Group 2: B Group 3: C A homologous rate of group assignment will be maintained. Neuropsychological assessment measurements and neurophysiological measures Neuropsychological assessment

To measure changes in the functioning of the cognitive processes of interest (Executive Functions, Attention, Memory and Social Cognition) we propose to use the following assessment instruments:

Neuropsychological Battery of Executive Functions and Frontal Lobes, 3rd Edition (BANFE-3)(Flores-Lázaro, et al. 2021). This is an instrument that allows exploring the functioning of 16 executive processes: Metamemory, figurative meaning comprehension, abstract attitude, verbal fluency, productivity, cognitive flexibility, visuospatial planning, sequential planning, inverse sequencing, encoding control, self-directed working memory, verbal working memory, visuospatial sequential working memory, inhibitory control, rule following and risk-benefit processing.

The exploration of these processes is performed through 14 tasks that were adapted from paradigms already tested in neuropsychological and neuroimaging studies in previous international studies. According to the authors, the test has sufficient convergent and clinical validity. The reliability assessed through inter-rater agreement is .80. The parameters were obtained from its application in a sample of Mexican participants without atypical functioning conditions.

The tests of interest for this study are described below:

Stroop Effect: It is considered an indicator of inhibitory control functioning since it evaluates the participant's ability to stop an automatic response and execute a non-dominant one. In this version, a sheet is used in which columns of six words are presented with color names that presuppose two conditions, in the neutral condition the person should only read the word that corresponds to the color of the ink with which it is printed on the sheet, while in the conflict condition, the participant must name the color of the ink with which the word is printed avoiding reading it, in this condition there is no concordance between the word and the color of the ink so that a situation of cognitive conflict is generated.

Card game: Adapted from the Iowa card test developed by Antoine Bechara (2003) and which explores the participant's ability to select a response under conditions of uncertainty and to detect risk-benefit relationships, so it is considered a sensitive task to measure decision making. The task is posed as a game in which the participant is presented with 10 decks of cards, five in which each one contains cards numbered from one to five respectively, and five that are placed in front of them and in which the cards are placed face down as they contain possible "punishments" that imply losing points. The task of the person being evaluated is to earn as many points as possible by choosing one card at a time from the five decks with the visible numbers. For each card selected, the evaluator will turn over one card from the corresponding deck to find out if it contains any punishment.

Tower of Hanoi: It is considered a sensitive task to evaluate the ability to plan sequential actions to achieve a specific goal. For its application, a toy is used that consists of a wooden base with three bars placed vertically at the same distance and a set of disks of different sizes that can be inserted into the bars. The activity consists of the participant moving the disks in order from smallest to largest size by placing them on the first bar towards the third bar following three main rules: no more than one disk can be moved at a time, larger disks cannot be placed on top of a smaller one, and the participant can only move one disk at a time.

placed on top of a smaller one and when removing them, they must always be placed on one of the bars. In this set there are two levels of difficulty according to the number of discs (three and four).

Alphabetical word order: According to the original authors of this paradigm, it evaluates the capacity to maintain information in working memory and manipulate it mentally. The participant must listen to a list of words and repeat it according to the alphabetical order of the initial. The list can be repeated in a maximum of five trials. Three lists are presented that progressively increase in complexity by number of words and by use of consonants and vowels.

Letter Sorting: This task is based on the Wisconsin letter sorting test and has been associated with cognitive flexibility functioning. Here the participant is asked to look at a base sheet containing the image of four cards that have geometric shapes that vary in shape, color, and number of shapes on each card. The participant is given a deck of 64 cards with the same characteristics and is asked to place each one of them under the card that he/she believes corresponds to the card on the sheet based on its characteristics. The evaluator can only answer yes or no according to a criterion established by the evaluator and that will change progressively but is not perceptible to the individual. The ability of the participant to modify his/her classification criterion according to the feedback provided by the evaluator is explored, especially in the conditions of criterion change.

Metamemory: This task evaluates the individual's ability to predict his own performance in a task of learning a list of words. The test consists of the subject trying to repeat a list of nine words in any order but trying to learn as many as possible over five trials. Before each trial, the participant must make a prediction of how many words he/she will be able to repeat, taking into consideration his/her performance in the previous repetitions and the perception he/she has of his/her own memory.

Behavioral assessment of executive function for adults (BRIEF-A) (Roth, Isquith & Gioia, 2005): this is a response inventory composed of 75 statements that are answered on a Likert scale with three options: never, sometimes and frequently. It yields results grouped into nine clinical scales: inhibition, flexibility, emotional control, self-monitoring, initiative, working memory, planning/organization, task monitoring and organization of materials, and three composite indices: Emotional Regulation Index, Metamemory Index, and Global Composite of Executive Functioning. It also offers three validity scales: denial, infrequency and inconsistency. This test does not have norms for Mexican population but it has been widely used in the context of research in Mexico and Latin America because it allows evaluating executive functioning in an ecological way.

NEUROPSI Attention and Memory 3 ed (Ostrosky et al. 2019). It is a neuropsychological assessment instrument that includes the assessment of three cognitive domains: Attention, Memory and Executive Functioning through tasks of different level of complexity and different sensory modalities. It evaluates people between 6 and 85 years old and its norms are based on Mexican population. According to the authors of the test, it has an adequate sensitivity to detect clinical alterations, so it is considered to have appropriate levels of discriminatory validity.

For the present project we intend to implement tasks to determine changes in attention and memory processes. The tasks are described below:

Digit retention in progression: this is a classic task to assess attention in the auditory modality. It consists of the presentation of numerical sequences of increasing length that the participant must repeat in the same order in which they were presented.

Digit detection: This is a task to assess attention. The participant must listen to a series of numbers numbers while they are read by the evaluator and when he/she hears the number 5 preceded by the number 2, he/she must tap the table.

Memory curve: This task consists of the participant having to listen to a list of 12 words during three consecutive repetitions, after each of which he/she must try to retrieve as many words as possible, regardless of the order in which they are repeated. For the evocation phase, after 30 minutes, the patient will be asked to try to spontaneously retrieve as many words as possible.

Gaze test: This test was originally designed in 2001 by Baron-Cohen with the aim of assessing the ability of individuals to detect intentions through facial expressions focused on the gaze. The computerized version developed by Galindo et al. (2018) will be used, which consists of 28 trials in which visual stimuli are presented showing the eyes of people making a particular expression that the participant must identify by selecting from four possible options. This instrument will be used to assess social cognition functions.

Neurophysiological recording Instruments and materials A resting-state electroencephalography neurophysiological recording of each participant will be performed in an artifact-free room using a 14-channel Emotiv EPOC. The datasets will be stored in the research mainframe for subsequent property extraction and offline analysis using artificial intelligence tools and techniques.

Stage 2. Intervention The interventions will be carried out through a 9-week group training that will be composed of 14 sessions of 60 minutes, and will be administered twice a week, by a professional psychologist with experience in the application of Mindfulness and CBT techniques according to the corresponding group (ANNEX intervention programs).

Follow-up Intervention Self-assessment record of intervention findings (optional). Beck Anxiety Inventory.

For the measurement of depression, the Beck Hopelessness Scale is used, composed of 20 items and three factors validated in Mexican population by Quiñonez-Tapia et al (2019).

For the measurement of anxiety, the Beck anxiety scale composed of 21 items and four factors Subjective, Neurophysiological, Autonomic, Vasomotor symptoms, validated in Mexican population by Vázquez et al. (2015) is used.

Neuropsychological assessment measures and neurophysiological measures Stage 3. Blind 3. Statistical analysis The project statistician will perform the comparisons of the results of the groups in ignorance of the assignment of labels of each group, as well as free of the assignment of the participants to the same and will return to the principal investigator the results outputs. ANOVA will be applied for hypothesis testing.Technique and Sample size calculation.

The sample considered for the study is 125 participants,calculated for the comparison of means of five groups with 22 participants each, expecting an effect size of 0.4, probability of error type 0.05, a power (1-prob err) of 0.95.

ELIGIBILITY:
Inclusion Criteria:

* Young adults 18-30 years old
* University students enrolled in any of the Autonomous University of Baja California programs.
* To properly accomplish to all assessment procedures
* To properly accomplish at least 80% of the intervention sessions
* Interest to voluntarly participate.

Exclusion Criteria:

* Disgnosis of neurological or psychitric disease, including severe anxiety or depression.
* Incomplete protocol evaluation.
* Out of 18-30 years old range age.
* Being enrolled in a different psychological or psychiatric intervention or treatment program during the period of evaluation and intervention.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological measures | Pre-post intervention assessment, after 8 weeks. A follow-up measure will be recorded immidiatly after each intervention session, 8 weeks as well.
  Neurophysiological, electroencephalographic (EEG) recordings will be performed:
  Each participant will undergo a five minute EEG recording in resting state, previous to any intervention, 128 Hz sampling rate, from 8 ch, EMOTIV Epoc (AF3, AF4, F3, F4, F7, F8, FC5, FC6), with saline solution for conductivity improvement. Offline EEG features frontal alpha-beta proportion change (if any) will be calculated using windowing power spectra transform. Follow-up five minutes, recordings after each intervention session and post-intervention program will be performed as well.
Mood measures | Pre-post intervention assessment, after 8 weeks.
  Anxiety and depression index will be calculated from Beck's adapted and validated version to Mexican population. Scores range from 0 min-30 max, normal score ranges from 25-30.
Card Sorting Test | Pre-post intervention assessment, after 8 weeks.
  Card Sorting Test, will be measured from the standardized executive function test BANFE, using accurcy of response, perseverations, time, and errors. Total score is transformed to normalized points 0-19 (with a mean of 10 ±3 SD, 4-6 low, 14-19 high performance).
Self directed signaling | Pre-post intervention assessment, after 8 weeks.
  Self directed signaling, will be measured from the standardized executive function test BANFE, using accuracy of response, time, and errors. Total score is transformed to normalized points 0-19 (with a mean of 10 ±3 SD, 4-6 low, 14-19 high performance).
Stroop Test | Pre-post intervention assessment, after 8 weeks.
  Stroop test, will be measured from the standardized executive function test BANFE, using accuracy of response, stroop type error, no-Stroop errors, and time, Total score is transformed to normalized points 0-19 (with a mean of 10 ±3 SD, 4-6 low, 14-19 high performance).
Working memory | Pre-post intervention assessment, after 8 weeks.
  Working Memory will be measured from the standardized executive function test BANFE, using accuracy of response as scoring criteria. Total score is transformed to normalized points 0-19 (with a mean of 10 ±3 SD, 4-6 low, 14-19 high performance).
Gambling test | Pre-post intervention assessment, after 8 weeks.
  Gambling test, will be measured by calculating EF quotients from the standardized test BANFE using risk cards percentage, final total score. Total score is transformed to normalized points 0-19 (with a mean of 10 ±3 SD, 4-6 low, 14-19 high performance).
Tower of Hanoi | Pre-post intervention assessment, after 8 weeks.
  Tower of Hanoi, using number of movements, and time, will be measured by calculating EF quotients from the standardized test BANFE. Total score is transformed to normalized points 0-19 (with a mean of 10 ±3 SD, 4-6 low, 14-19 high performance).
Metamemory | Pre-post intervention assessment, after 8 weeks.
  Metamemory, will be measured by calculating EF quotients from the standardized test BANFE using positive and negative errors. Total score is transformed to normalized points 0-19 (with a mean of 10 ±3 SD, 4-6 low, 14-19 high performance).
Neuropsychological evaluation | Pre-post intervention assessment, after 8 weeks.
  Attention and Memory, normilized quotient will be calculated according to NEUROPSI standard Attention and Memory Standardized test, using accuracy of response, and time as direct measures of each task. Attention and memory score is normalized according to age and years of education, scores range from 1-19 (1-3 extremely low, 4-6 low, 7-13 normal, 14-19 high performance).
Neuropsychological measure | Pre-post intervention assessment, after 8 weeks.
  Social Cognition, according to index from computarized adapted version of the Mind in the Eyes test, index 0 (min) - 36 (max) score, expected score ranges from 25-36.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Autónoma de Baja California, Neuroscience and Cognition Laboratory, Mexicali, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No
No need for IPD sharing in this protocol, the interventions are preventive order, and the evaluations are intended to identify survival for protective cognitive features, no medical conditions issued.